CLINICAL TRIAL: NCT05578053
Title: Efficacy and Safety of Dalpiciclib in Hormone Receptor-positive Advanced Breast Cancer: a Multicenter, Observational, Real-world Study
Brief Title: Efficacy and Safety of Dalpiciclib in Hormone Receptor-positive Advanced Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Cuizhi GENG, Vice President of Hebei Medical University Fourth Hospital, Hebei Medical University Fourth Hospital
Other Study IDs: 2022106
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- locally advanced/metastatic HR+ breast cancer patients: HR+ postmenopausal or premenopausal and locally advanced or metastatic breast cancer patients who had received or had not received prior systemic therapy.
  Interventions: Drug: Dalpiciclib

INTERVENTIONS:
Drug: Dalpiciclib — a new, orally administered, selective CDK4/6 inhibitor
  Other Names: SHR-6390

SUMMARY:
This study is a multi-center, observational, real-world study. We planned to recruit 420 HR+ locally advanced or metastatic breast cancer patients who had received or had not received prior systemic therapy. All patients included in the analysis were receiving or planning to receive dalpiciclib-containing regimens without restrictions, completely following the physician 's clinical choice, to assess the efficacy and safety of dalpiciclib-containing regimens.

DETAILED DESCRIPTION:
All patients included in the analysis were receiving or were planning to receive dalpiciclib and other standard therapy, with no restrictions on the regimen and full adherence to physician clinical choices. Patients who qualified after completing the screening tests and assessments entered the study treatment period and were treated and visited with a dalpiciclib -containing regimen as specified in the protocol. Patients underwent imaging assessments and safety assessments according to clinical routine during study treatment, with the investigator 's assessment as the final result.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years, postmenopausal or premenopausal female or male patients, female patients must meet one of the following: a) previous bilateral oophorectomy, or age ≥ 60 years; b) age < 60, natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH at postmenopausal levels; c) premenopausal or perimenopausal female patients can also be enrolled, but must be willing to receive LHRH agonist therapy during the study;
2. pathological examination confirmed HR-positive male/female breast cancer patients, with evidence of focal recurrence or metastasis, not suitable for surgical resection or radiation therapy with the purpose of cure;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
4. Serum pregnancy test must be performed within 28 days before enrollment in women of childbearing age and the result is negative,And male/female patients are willing to use a medically recognized highly effective contraceptive during the study and within 1 year after the last dose of study drug;
5. non-pregnant or non-lactating female patients；
6. do not participate in other ongoing studies at the same time ；
7. agreed by the patient himself or her legal representative and have signed an informed consent form, willing and able to comply with scheduled visits, study treatment plan, laboratory tests and other trial procedures.

Exclusion Criteria:

1. any evidence of serious or uncontrolled systemic disease, including uncontrolled hypertension, active bleeding disorders, active infections, including hepatitis B, C, and human immunodeficiency virus, or severely impaired bone marrow reserve or organ function, including liver and kidney damage, which, in the opinion of the investigator, would greatly alter the balance of wind benefit/risk.
2. at the time of initiation of dalpiciclib treatment, the patient has not recovered from any CTCAE grade ≥ 3 toxicity caused by previous treatment
3. known history of hypersensitivity to dalpiciclib or excipients or drugs with similar chemical structure to dalpiciclib
4. patients who are considered unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+ postmenopausal/premenopausal locally advanced/metastatic breast cancer patients who had received or had not received prior systemic therapy were planned to be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  progression free survival
AE | 2 years
  the incidence of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Cuizhi Geng Cuizhi Geng, archiater, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth hospital of Hebei University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided